CLINICAL TRIAL: NCT04165616
Title: MECHANIST: Motor rECovery witH eArly imagiNg In STroke
Brief Title: Motor rECovery witH eArly imagiNg In STroke
Acronym: MECHANIST
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Julius Dewald, Professor and Chair, Northwestern University
Other Study IDs: STU00210349; R01NS105759 (NIH)
Record Dates: First submitted 2019-10-30; First posted 2019-11-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with stroke

SUMMARY:
This study will contribute to the field of stroke rehabilitation research by expanding the investigator's understanding of the neural mechanisms responsible for the development and expression of abnormal flexion synergy, a primary movement impairment due to stroke. The study will longitudinally evaluate motor tract morphology and motor impairment/function in an attempt to develop early neuroimaging-based predictors of the development of flexion synergy and its impact on reaching and hand recovery (6 month). The study will utilize quantitative motor testing (kinematics and kinetics) to measure motor impairment and reaching and hand function. Both neuroimaging and quantitative motor testing will be conducted within 96 hours-, 2 weeks-, 3 months-, and 6 months-post stroke. The knowledge gained by this study will provide crucial structural and functional neuroimaging evidence that demonstrates the timeline of progressive ipsi- and contralesional motor pathway (including bulbospinal pathways) changes and the associated development of flexion synergy that grossly impacts reaching and hand function in individuals with moderate to severe stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke within the middle cerebral artery distribution based on brain MRI done within 48 hours of admission
2. 18 to 85 years old
3. Isolated motor deficits (hemiparesis) without significant aphasia, visual disturbances, or neglect based on the following scores on the NIH Stroke Scale: 1a (level of consciousness) = 0- Alert; keenly responsive. 1b (LOC questions) = 0- Asked month and age; Answers both correctly. 1c (LOC commands) = 0- Asked to open/close eyes, grasp/release hand; Performs both correctly. 2 (Best Gaze) = 0- Horizontal eye movements; Normal. 5 (Motor Arm) = 1, 2, 3, or 4- Arm placed at 90 (sitting) or 45 (supine), Drift, Some effort, No effort against gravity, or No movement. 7 (Limb Ataxia) = 0- Finger-nose-finger or heel-shin test; Absent. 8 (Sensory) = 0 or 1- Pin prick; Normal or Mild-to-moderate sensory loss. 9 (Best Language) = 0 or 1- Describe picture; No or Mild-to-moderate Aphasia. 11 (Extinction and Inattention) = 0 or 1- No abnormality or Inattention to one modality.

Exclusion Criteria:

1. Premorbid disability or sensorimotor impairment
2. Comorbidity medically contraindicating the administration of subsequent MRI scanning and motor assessments
3. Pain or hypersensitivity limiting motor assessment
4. Limb edema limiting motor assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the in-patient stroke unit based upon the study inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in fractional anisotropy | Change in fractional anisotropy will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Fractional anisotropy is a quantitative measure of fiber density, axonal diameter, and myelination in the corticofugal, corticoreticulospinal, and corticorubrospinal tracts derived from the diffusion tensor imaging dataset.
Change in complexity | Change in complexity will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Complexity (alpha) is an index of the non-Gaussian diffusion dynamics within the corticofugal, corticoreticulospinal, and corticorubrospinal tracts derived from the diffusion tensor imaging dataset.
Change in mean diffusivity | Change in mean diffusivity will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Mean diffusivity is a measure of neural tract integrity quantifying the rotationally invariant magnitude of water diffusion within neural tissue defined by the 3-dimensional diffusion tensor.
Change in radial diffusivity | Change in radial diffusivity will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Radial diffusivity is a measure of neural membrane integrity quantifying the average of the two small-axis values of water diffusion within neural tissue defined by the 3-dimensional diffusion tensor.
Change in axial diffusivity | Change in axial diffusivity will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Axial diffusivity is a measure of neural tract direction quantifying the long-axis value of water diffusion within neural tissue defined by the 3-dimensional diffusion tensor.
Change in maximum reaching distance | Change in maximum reaching distance will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Quantitative evaluation of reaching accounting for the expression of both flexion synergy and weakness by calculating distance from reaching kinematics data during ballistic outward reaches against various abduction loads.
Change in maximum hand aperture | Change in maximum hand aperture will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Quantitative evaluation of hand opening accounting for the expression of both flexion synergy and weakness by calculating the area of a pentagon formed by the finger tips from hand kinematics data obtained at various abduction loads.
Change in maximum grasp force | Change in maximum grasp force will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Quantitative evaluation of hand closing accounting for the expression of both flexion synergy and weakness by calculating the mean surface grasp force of the hand at various abduction loads.
Predictive capacity of diffusor tensor imaging (DTI) for 6-month reaching and hand performance | Changes in structural morphology from 48 hours to 2-weeks post-stroke will be evaluated as early predictors for the 6-month reaching and hand performance outcomes including ROC curve analysis.
  Changes in structural morphology measured acutely will be evaluated as early predictors for chronic reaching and hand performance. Receiver operating characteristic (ROC) curve analysis will be used to evaluate the discrimination potential of each acute imaging measure in predicting chronic moderate versus severe motor impairment for each of the reaching and hand performance measures.
Relationship between DTI and quantitative motor testing | Relationships between metrics will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  The relationship between each structural morphology metric and each quantitative motor testing metric will be evaluated.

SECONDARY OUTCOMES:
Change in Fugl-Meyer Motor Assessment | Change in Fugl-Meyer Motor Assessment will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Qualitative and clinical assessment of general motor impairment of arm following stroke. The scale evaluates movement impairment of the arm through observation. The scale ranges from 0-66 points with 66 indicating the best score.
Change in Action Research Arm Test | Change in Action Research Arm Test will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Qualitative and clinical assessment of activity limitation (function) of the arm following stroke. The scale focusses on reaching, grasping, and releasing objects of various sizes. The scale ranges from 0-57 with 57 indicating the best score.
Change in Stroke Impact Scale | Change in Stroke Impact Scale will be modeled over 4 time points (48-96 hours-, 2 weeks-, 3 months-, and 6 months post-stroke).
  Structured interview to assess domains of the ICF (International Classification of Functioning, Disability and Health) in individuals following stroke. The domains include self-reported physical problems, memory and thinking, control of emotions, communication, daily activities, home and community mobility, the affected hand, participation and life roles, and global recovery. Each domain score is transformed to a scale of 0-100 with 100 being the best score.

CONTACTS AND LOCATIONS:
Overall Officials: Julius PA Dewald, PT, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Department of Physical Therapy and Human Movement Sciences, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Shirley Ryan AbilityLab, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Final research data will be shared openly and timely in accordance with NIH Data Sharing Policy (https://grants.nih.gov/grants/policy/data_sharing/). Data sharing will occur through the primary repositories of Northwestern University DigitalHub (https://prism.northwestern.edu/) and Open Science Framework (https://osf.io/). Data will be exported from the internal RedCap study data base in spreadsheet format and will be deidentified and coded. Data will be available through speaking engagements and publications, presentations at scientific symposia and seminars. Data sharing in the above repositories will be phased in time with acceptance for publication of the primary outcome paper near the end of the fifth year and then with each subsequent publication. Publications will include DOIs for the data repositories.
Time Frame: Data sharing in the above repositories will be phased in time with acceptance for publication of the primary outcome paper near the end of the fifth year and then with each subsequent publication.
Access Criteria: Data sharing will occur through the primary repositories of Northwestern University DigitalHub (https://prism.northwestern.edu/) and Open Science Framework (https://osf.io/). Data will be exported from the internal RedCap study data base in spreadsheet format and will be deidentified and coded.
URL: https://prism.northwestern.edu/

REFERENCES:
- [Background] Karbasforoushan H, Cohen-Adad J, Dewald JPA. Brainstem and spinal cord MRI identifies altered sensorimotor pathways post-stroke. Nat Commun. 2019 Aug 6;10(1):3524. doi: 10.1038/s41467-019-11244-3. PMID 31388003
- [Background] McPherson JG, Chen A, Ellis MD, Yao J, Heckman CJ, Dewald JPA. Progressive recruitment of contralesional cortico-reticulospinal pathways drives motor impairment post stroke. J Physiol. 2018 Apr 1;596(7):1211-1225. doi: 10.1113/JP274968. Epub 2018 Feb 19. PMID 29457651
- [Background] Yamada K. The glossophyaryngeal nerve response to taste and thermal stimuli in the rat, rabbit and cat. Kumamoto Med J. 1965 Jun 30;18(2):106-8. No abstract available. PMID 5825888